CLINICAL TRIAL: NCT00186550
Title: An Evaluation of Group Psychotherapy for People With HIV
Brief Title: Group Psychotherapy for People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Spiegel, Jack, Lulu & Sam Willson Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH054930-04 (NIH); R01MH054930-04 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: HIV; Depression; Risk-taking; Pain
MeSH Terms: conditions — Depression; Risk-Taking; Pain | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Supportive Expressive Group Psychotherapy
Behavioral: Education

SUMMARY:
This study will examine the effectiveness of supportive-expressive group therapy plus education compared with an educational intervention in improving the quality of life and promoting health-enhancing behavior of men and women living with HIV or AIDS.

DETAILED DESCRIPTION:
The major goal of this project is to examine the effectiveness of supportive-expressive group therapy plus education in comparison to an educationally intervention in improving the quality of life and promoting health-enhancing behavior of men and women living with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* 1) a positive HIV diagnosis (either symptomatic or asymptomatic), 2) at least eighteen years of age, 3) English language skill (to complete questionnaires and participate, if assigned, to the group psychotherapy condition) and, 4) geographical proximity to groups in order to attend if assigned.

Exclusion Criteria:

* 1) severe psychiatric disorders (i.e. schizophrenia or other psychotic disorders)who would not be appropriate for participating in the group intervention, 2) active tuberculosis, 3) acute intoxication, 4) participation in an ongoing HIV/AIDS support group or 5) suicidal/homicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Power R, Gore-Felton C, Vosvick M, Israelski DM, Spiegel D. HIV: effectiveness of complementary and alternative medicine. Prim Care. 2002 Jun;29(2):361-78. doi: 10.1016/s0095-4543(01)00013-6. PMID 12391716
- [Result] Vosvick M, Gore-Felton C, Ashton E, Koopman C, Fluery T, Israelski D, Spiegel D. Sleep disturbances among HIV-positive adults: the role of pain, stress, and social support. J Psychosom Res. 2004 Nov;57(5):459-63. doi: 10.1016/j.jpsychores.2004.03.003. PMID 15581649
- [Result] Gore-Felton C, Vosvick M, Bendel T, Koopman C, Das B, Israelski D, Herrera M, Litzenberg K, Spiegel D. Correlates of sexually transmitted disease infection among adults living with HIV. Int J STD AIDS. 2003 Aug;14(8):539-46. doi: 10.1258/095646203767869156. PMID 12935384
- [Result] Power R, Koopman C, Volk J, Israelski DM, Stone L, Chesney MA, Spiegel D. Social support, substance use, and denial in relationship to antiretroviral treatment adherence among HIV-infected persons. AIDS Patient Care STDS. 2003 May;17(5):245-52. doi: 10.1089/108729103321655890. PMID 12816618
- [Result] Gore-Felton C, Vosvick M, Power R, Koopman C, Ashton E, Bachmann MH, Israelski D, Spiegel D. Alternative therapies: a common practice among men and women living with HIV. J Assoc Nurses AIDS Care. 2003 May-Jun;14(3):17-27. doi: 10.1177/1055329003014003002. PMID 12800809
- [Result] Koopman C, Gore-Felton C, Azimi N, O'Shea K, Ashton E, Power R, De Maria S, Israelski D, Spiegel D. Acute stress reactions to recent life events among women and men living with HIV/AIDS. Int J Psychiatry Med. 2002;32(4):361-78. doi: 10.2190/CK2N-33NV-3PVF-GLVR. PMID 12779186
- [Result] Vosvick M, Koopman C, Gore-Felton C, Thoresen C, Krumboltz J, Spiegel D. Relationship of functional quality of life to strategies for coping with the stress of living with HIV/AIDS. Psychosomatics. 2003 Jan-Feb;44(1):51-8. doi: 10.1176/appi.psy.44.1.51. PMID 12515838
- [Result] Turner-Cobb JM, Gore-Felton C, Marouf F, Koopman C, Kim P, Israelski D, Spiegel D. Coping, social support, and attachment style as psychosocial correlates of adjustment in men and women with HIV/AIDS. J Behav Med. 2002 Aug;25(4):337-53. doi: 10.1023/a:1015814431481. PMID 12136496
- [Result] Koopman C, Gore-Felton C, Marouf F, Butler LD, Field N, Gill M, Chen XH, Israelski D, Spiegel D. Relationships of perceived stress to coping, attachment and social support among HIV-positive persons. AIDS Care. 2000 Oct;12(5):663-72. doi: 10.1080/095401200750003833. PMID 11218551
- [Result] Gore-Felton C, Butler LD, Koopman C. HIV disease, violence, and post-traumatic stress. Focus. 2001 May;16(6):5-6. No abstract available. PMID 11547387